CLINICAL TRIAL: NCT03659344
Title: Vicryl Plus and Vicryl Sutures in Reduce of Infection in Dental Implant Surgery
Brief Title: Efficacy of Antimicrobial Coating Suture Coated Vicryl Plus Compared With Vicryl in Reduced Surgical Site Infection of Dental Implant Surgeries: A Uni-Blind Randomized Clinical Trial Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, Associate professor of OMFS, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IR.SBMU.RIDS.REC.1395.336
Record Dates: First submitted 2018-08-31; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Infection, Surgical Site
Keywords: sutures; Surgical Wound Infection; Polyglactin 910
MeSH Terms: conditions — Surgical Wound Infection | interventions — Polyglactin 910

STUDY DESIGN:
Intervention Model Description: In group1, vicryl plus suture was used to close flaps. In group2,vicryl was used to close flaps
Who Masked: Participant
Masking Description: Patients were blind about kind of sutures which were used to close flaps.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl plus (Active Comparator): In this group, vicryl plus(Triclosan coated) sutures were used to close flaps
  Interventions: Drug: Vicryl plus
- vicryl (No Intervention): In this group, vicryl sutures were used to close flaps

INTERVENTIONS:
Drug: Vicryl plus — Using vicryl sutures which coated with triclosan (antibiotic)
  Arms: Vicryl plus

SUMMARY:
Patients randomly aligned in 2 groups.Vicryl plus sutures were used in group 1 for closing subperiostal flaps after dental implant surgeries and vicryl sutures were used in group 2.

DETAILED DESCRIPTION:
Patients were divided randomly based on computer randomization list in two groups: In group1, vicryl plus 4-0 (Vicryl Plus Ethicon,Johnson & Johnson Company, Sommerville, NJ) suture was used to close surgical site and Vicryl 4-0 (Vicryl Ethicon,Johnson & Johnson Company, Sommerville, NJ) in group II.

All dental implants were placed through creating subperiosteal flaps. In each group, fresh socket placed dental implants were documented. Patients were visited in 1, 2, 3 and 4 weeks after dental implant surgeries.

Postoperative infection was defined as local erythematous change in the sutured wound with purulent discharge or localized abscess formation on surgical site. If wound dehiscence occurred, it was documented.

Patients were blind about what suture was used.

ELIGIBILITY:
Inclusion Criteria:

* Need 3 dental implants at the posterior of the mandible

Exclusion Criteria:

* Diabetic patients
* smoker
* poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of post-operative infection | In one month
  The number of participants who had local erythematous change in the sutured wound with purulent discharge or localized abscess formation on surgical site.
The prevalence of post-operative dehiscence | In one month
  The number of participants who had relatively or completely open wound

IPD SHARING:
Plan to Share IPD: No